CLINICAL TRIAL: NCT07177651
Title: Comparative Study Between Laminoplasty Versus Laminectomy With Lateral Mass Fixation in Management of Degenerative Cervical Canal Stenosis
Brief Title: Laminoplasty Versus Laminectomy With Lateral Mass Fixation in Management of Degenerative Cervical Canal Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fahd Abdel Sabour Ahmed Mohammed, Principal investigator, specialist , neurosurgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Posterior cervical approaches
Record Dates: First submitted 2025-07-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Stenosis; Degenerative Cervical Spinal Stenosis
Keywords: Laminoplasty; Lateral mass fixation
MeSH Terms: interventions — Laminoplasty; Laminectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laminoplasty (Experimental)
  Interventions: Procedure: Laminoplasty
- Laminectomy with lateral mass fixation (Experimental)
  Interventions: Procedure: Laminectomy with lateral mass fixation

INTERVENTIONS:
Procedure: Laminoplasty — Is a posterior approach that involves the surgical widening of the spinal canal by reshaping or repositioning the lamina. However, some patients with cervical stenosis
  Arms: Laminoplasty
Procedure: Laminectomy with lateral mass fixation — Posterior cervical decompression with lateral mass screw insertion
  Arms: Laminectomy with lateral mass fixation

SUMMARY:
Cervical canal stenosis (CCS) is a condition characterized by the narrowing of the spinal canal in the cervical spine, leading to compression of the spinal cord and nerve roots. This can result in a variety of neurological deficits, including myelopathy, radiculopathy, and motor dysfunction. The primary goal of treatment is to relieve neural compression and improve or preserve neurological function. Surgical decompression, such as laminoplasty, is a common procedure to treat this condition, as it decompresses the spinal canal to relieve pressure on the spinal cord. Laminectomy with lateral mass fixation is another option of management.

DETAILED DESCRIPTION:
Cervical canal stenosis (CCS) is a condition characterized by the narrowing of the spinal canal in the cervical spine, leading to compression of the spinal cord and nerve roots. This can result in a variety of neurological deficits, including myelopathy, radiculopathy, and motor dysfunction. The primary goal of treatment is to relieve neural compression and improve or preserve neurological function. Surgical decompression, such as laminoplasty, is a common procedure to treat this condition, as it decompresses the spinal canal to relieve pressure on the spinal cord.

Laminoplasty is a posterior approach that involves the surgical widening of the spinal canal by reshaping or repositioning the lamina. However, some patients with cervical stenosis, particularly those with accompanying spinal instability or degenerative changes, may not achieve satisfactory outcomes with laminoplasty alone. In such cases, lateral mass fixation is often added to provide supplemental stability to the spine, potentially preventing postoperative deformities and enhancing long-term outcomes

Lateral mass fixation is often combined with posterior decompression and typically done as part of a posterior cervical fusion where screws are placed into the lateral masses (bony structures on the sides of the vertebrae) to stabilize the cervical spine after decompression, such as through a laminectomy. This procedure sacrifices some motion for stability.

A comparative study is needed to better understand the advantages and disadvantages of each approach, in order to guide clinical decision-making and improve patient outcomes.

The general aim is to evaluate and compare the clinical outcomes, safety, and effectiveness of both surgical techniques in managing this condition.

The specific aim is to compare the clinical efficacy, assess the radiological outcomes, evaluate the surgical and postoperative complication and investigate long-term outcomes and instability.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 ≥ years with clinically significant cervical canal stenosis (based on imaging and neurological symptoms).
* Surgical indication for cervical decompression.
* Adequate follow up data (minimum 1 year).
* Patients fit for surgery.

Exclusion Criteria:

* Patients unfit for surgery or contraindication to general anaesthesia.
* Congenital deformities or significant spinal deformities unrelated to stenosis.
* Patients with cervical kyphosis, active infection or known allergy to titanium.
* Previous cervical spine surgery.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-10-04 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in modified Japanese Orthopaedic Association (mJOA) score from baseline to 6 months (neurological function; range 0-17; higher = better function) | Baseline and 6 months postoperatively
  Neurological outcome will be assessed using the modified Japanese Orthopaedic Association (mJOA) score, which evaluates motor and sensory function of the upper and lower extremities, as well as bladder function. Scores range from 0-17, with higher scores indicating better neurological function. Assessments will be performed at baseline (pre-operative), and at 6 months postoperatively by a blinded clinician.

SECONDARY OUTCOMES:
Complication rate within 90 days postoperatively | Within 90 days postoperatively
  All perioperative complications will be recorded within 90 days of surgery, including but not limited to surgical site infection (CDC criteria), C5 palsy (new postoperative motor deficit in deltoid/biceps), cerebrospinal fluid leak, and reoperation for any cause.
Length of hospital stay (days) | Perioperative period
  Length of hospital stay will be recorded as the number of days from surgery to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Hassan Ragab, Study Director — Assiut University hospital, neurosurgery department; Abdel Hakeem Abdel Sattar, Study Director — Assiut University, neurosurgery department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] https://www.asianspinejournal.org/journal/view.php?doi=10.4184%2Fasj.2016.10.3.536
- See also: Related Info — https://www.nature.com/articles/3101477